CLINICAL TRIAL: NCT02520167
Title: Partnership to Improve Nutrition and Adiposity in Prenatal Clinical Care: a Pilot and Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Denver Health and Hospital Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15-0760
Record Dates: First submitted 2015-08-05; First posted 2015-08-11 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Pregnancy
Keywords: Gestational weight gain
MeSH Terms: conditions — Gestational Weight Gain | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary and Lifestyle Counseling (Experimental): Women randomized to the intervention group will meet with a dietary counselor for 15 minutes at every prenatal appointment. They will receive a dietary and lifestyle curriculum based on the Diabetes Prevention Program curriculum (11 lessons) with one additional lesson providing prenatal breastfeeding education. They will also have access to a private online Facebook page for additional education and peer group support.
  Interventions: Behavioral: Dietary and Lifestyle Counseling
- Standard of Care (No Intervention): Usual prenatal care consists of regular clinical appointments, pregnancy ultrasounds, and recommendations to use prenatal multivitamins, eat a balanced diet, and remain physically active. Women with a pre-pregnant body mass index > 30 complete early glucose screening (as early as possible after presentation at the clinic) to detect pre-existing diabetes, and all women undergo routine gestational diabetes screening at 24-28 weeks. Women who test positive for pre-existing diabetes or gestational diabetes are referred to a registered dietitian.

INTERVENTIONS:
Behavioral: Dietary and Lifestyle Counseling — Dietary and lifestyle education; Peer group support.
  Arms: Dietary and Lifestyle Counseling

SUMMARY:
This study will pilot and assess feasibility of a prenatal intervention for obese pregnant women based on the Diabetes Prevention Program (DPP). Intervention group participants will meet with a clinic dietitian for 15 minutes at every prenatal appointment to complete a DPP-based curriculum and receive breastfeeding education. Control group participants will receive usual prenatal care. Outcomes include reach and dose of the intervention, gestational weight gain, dietary intake, physical activity, and breastfeeding in the first 6 weeks postpartum.

DETAILED DESCRIPTION:
This study will pilot and test feasibility of a prenatal lifestyle intervention designed to limit gestational weight gain and prevent gestational diabetes. The intervention is based on the Diabetes Prevention Program lifestyle intervention, will include prenatal breastfeeding education and online peer group support, and will be integrated into the participants' regular prenatal appointments. Women (n=24) will be enrolled in early pregnancy. After baseline assessments (demographics, maternal diet, physical activity, mental health), women randomized equally to the intervention or usual care conditions. Further data collection will occur at approximately 24 weeks gestation, 36 weeks gestation, and 6 weeks postpartum, and clinical data (weight, pregnancy and obstetric complications) will be abstracted from medical records at the end of the study. Outcomes include reach and dose of the intervention, gestational weight gain, dietary intake, physical activity, and breastfeeding in the first 6 weeks postpartum. The investigators hypothesize that the intervention will reduce gestational weight gain, improve maternal dietary intake, increase total energy expenditure, and increase breastfeeding exclusivity in the first 6 weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies of <12 weeks gestation
* Pre-pregnant body mass index >=30
* Speak and understand English
* Plan to continue care at the clinic through pregnancy and postpartum

Exclusion Criteria:

* Pre-existing diabetes
* History of serious chronic illnesses
* History of prior gestational diabetes
* Prior delivery at <37 weeks gestation
* Prior delivery of infant weighing <2500g

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain | 40 weeks
  Weight change from pre-pregnancy to time of delivery

SECONDARY OUTCOMES:
Maternal fruit intake | Assessed from 12 weeks gestation through 6 weeks postpartum
  Change in daily servings of fruit from early pregnancy to mid-pregnancy, late pregnancy, and postpartum
Maternal vegetable intake | Assessed from 12 weeks gestation through 6 weeks postpartum
  Change in daily servings of vegetables from early pregnancy to mid-pregnancy, late pregnancy, and postpartum
Maternal whole grains intake | Assessed from 12 weeks gestation through 6 weeks postpartum
  Change in daily servings of whole grains from early pregnancy to mid-pregnancy, late pregnancy, and postpartum
Maternal solid fats intake | Assessed from 12 weeks gestation through 6 weeks postpartum
  Change in daily servings of solid fats from early pregnancy to mid-pregnancy, late pregnancy, and postpartum
Maternal added sugars intake | Assessed from 12 weeks gestation through 6 weeks postpartum
  Change in daily servings of added sugars from early pregnancy to mid-pregnancy, late pregnancy, and postpartum
Maternal physical activity | Assessed from 12 weeks gestation through 6 weeks postpartum
  Change in total estimated energy expenditure from early pregnancy to mid-pregnancy, late pregnancy, and postpartum
Exclusive breastfeeding | Assessed at 6 weeks postpartum
  Measured as exclusive breastfeeding (no formula, no complementary foods) in the first 6 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Sauder, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Denver Health Eastside Family Health Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available for this small pilot and feasibility study